CLINICAL TRIAL: NCT02086565
Title: Using IT to Improve Access, Communication and Asthma in African American and Hispanic/Latino Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R-1307-05218
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Results first posted 2019-06-05 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Asthma; Communication
Keywords: asthma,; asthma control,; asthma-related quality of life; electronic health record,; portal,; health literacy
MeSH Terms: conditions — Asthma; Communication | interventions — House Calls

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Portal training and home visits (Experimental): Portal training and home visits from a community health worker to promote care coordination and use of the patient portal
  Interventions: Behavioral: Portal training and home visits
- portal training (Active Comparator): Participants are assured internet access and taught to use the patient portal
  Interventions: Behavioral: Portal training

INTERVENTIONS:
Behavioral: Portal training and home visits — patient portal training and home visits by CHW to coordinate care
  Arms: Portal training and home visits
Behavioral: Portal training — training in use of patient portal
  Arms: portal training

SUMMARY:
Background: Asthma morbidity is high in inner-city minority adults, despite the existence of efficacious therapy. Tailored, patient-centered interventions are needed to improve access to care and patient-provider communication. Access and communication increasingly rely on information technology (IT) as new incentives arise to use the Electronic Health Record (EHR). The EHR patient portal (PP) gives patients web-based communication with providers and practices. How the poor and those with limited educational opportunities can take advantage of these is unclear. In contrast, the investigators have found that home visits (HVs) by community health workers (CHWs) can improve access to care for children and promote caretaker-clinician communication. The investigators also found many inner-city adults have internet access and are willing to learn to use the PP.

Objective: to examine the benefits for adults of using the PP with and without HVs by CHWs who will encourage/facilitate PP use, understand patients' social context, and enhance communication with the medical team. The investigator hypothesize all patients will benefit from PPs, and that the addition of HVs will be particularly helpful for those with low literacy or language barriers. Specific Aims test if the 1-year interventions result in 1) better within-group asthma outcomes, 2) better outcomes in one group over the other, 3) more communication (use of PP) and access (appointments made and kept) which mediate the interventions' effects on asthma outcomes, and 4) effect modification by literacy level, primary language, and convenience of internet access.

Methods: In a randomized controlled trial, 301 adults, predominantly African American and Hispanic/Latino, with uncontrolled asthma recruited from low income urban neighborhoods will be assured internet access and taught to use the PP, with and without HVs from a CHW. CHWs will 1) train patients to competency in PP use, 2) enhance care coordination, 3) transmit a view of the complex social circumstances of patients' lives to providers, and 4) make up for differences in patients' health literacy skills.

Patient Outcomes are asthma control, asthma-related quality of life, emergency department (ED) visits, and hospitalizations for asthma or any cause. Together asthma and other health conditions affect patients' ability to perform their daily tasks and care for their families. Potential benefits of the intervention are enhanced patient-clinician communication, access to care, improved health, and ability to use IT.

ELIGIBILITY:
Inclusion Criteria:

* adults predominantly African American and Hispanic/Latino with uncontrolled asthma recruited from low income urban neighborhoods

Exclusion Criteria:

* severe psychiatric or cognitive problems that would make it impossible to understand and complete the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2014-07-17 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea J Apter, MD, MSc, MA, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Localio AM, Klusaritz H, Morales KH, Ruggieri DG, Han X, Apter AJ. Primary language and the electronic health record patient portal: Barriers to use among Spanish-speaking adults with asthma. J Asthma. 2022 Oct;59(10):2081-2090. doi: 10.1080/02770903.2021.1989462. Epub 2021 Oct 20. PMID 34634975
- [Derived] Apter AJ, Localio AR, Morales KH, Han X, Perez L, Mullen AN, Rogers M, Klusaritz H, Howell JT, Canales MN, Bryant-Stephens T. Home visits for uncontrolled asthma among low-income adults with patient portal access. J Allergy Clin Immunol. 2019 Sep;144(3):846-853.e11. doi: 10.1016/j.jaci.2019.05.030. Epub 2019 Jun 7. PMID 31181221
- See also: Patient Centered Outcomes Research Institute — http://www.pcori.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We intended to enroll 300 participants. Because several research coordinators were working at once, and calls were pending to patients, we identified and enrolled and randomized 301 participants..
Period: Overall Study
Arm/Group | Portal Training and Home Visits | Portal Training
Started | 151 | 150
Completed | 135 | 138
Not Completed | 16 | 12
Not completed — Lost to Follow-up | 9 | 7
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Death | 3 | 2
Not completed — withdrawn by research team | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Portal Training and Home Visits | Portal Training | Total
Number analyzed (Participants) | 151 | 150 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (14) | 48 (12) | 49 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 134 | 270
  Male | 15 | 16 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 35 | 66
  Not Hispanic or Latino | 117 | 114 | 231
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 116 | 113 | 229
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 22 | 26 | 48
asthma control questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Asthma Control Questionnaire is a validated 6-item questionnaire, range 0 to 6, that reflects asthma symptoms over the past week. Lower score is better control.
  units on a scale | 2.4 (1.1) | 2.4 (1.2) | 2.4 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Score of Asthma Control Questionnaire
Description: This is a validated test with 6 items each with Likert score 0 to 6, reflecting symptoms over the past week. Lower score is a better outcome. We measured change in Asthma Control Questionnaire score from baseline to at least 12 months.
Time Frame: baseline and over a year
Population: The result is the mean change in asthma control (lower is improved control) at 12 months from baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Portal Training and Home Visits | Portal Training
Number analyzed (Participants) | 151 | 150
score on a scale | -0.48 [-0.76 to -0.22] | -0.27 [-0.52 to -0.01]
Statistical Analysis 1: Comparison: Portal Training and Home Visits vs Portal Training; Test type: Superiority; Group differences in expected 12 month c = -0.21, 95% CI 2-sided [-0.56 to 0.15]

2. Secondary Outcome: Asthma-related Quality of Life
Description: Quality of life is a 15-item questionnaire with 7 point response scale (1-7), higher score is better quality of life. We measured the change from baseline and over a year.
Time Frame: baseline and over a year
Population: Quality of life is a 15-item questionnaire with 7 point response scale (1-7), higher score is better quality of life. Here we measure change in quality of life over time in the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Portal Training and Home Visits | Portal Training
Number analyzed (Participants) | 151 | 150
score on a scale | 0.64 [0.31 to 0.98] | 0.45 [0.13 to 0.78]
Statistical Analysis 1: Comparison: Portal Training and Home Visits vs Portal Training; Test type: Superiority; Group differences in expected 12 month c = 0.19, 95% CI 2-sided [-0.27 to 0.68] — Estimation parameter: Other. Group differences in expected 12 month change from baseline

3. Secondary Outcome: Emergency Department Visits
Description: Emergency department visits for asthma from one year before baseline to one year after baseline.
Time Frame: one year before baseline to one year after baseline
Population: ED visits per year over period of participation
Measure: Least Squares Mean (95% Confidence Interval); unit: ED visits per year
Arm/Group | Portal Training and Home Visits | Portal Training
Number analyzed (Participants) | 151 | 150
ED visits per year | -3.29 [-4.73 to -2.10] | -2.69 [-3.67 to -1.88]
Statistical Analysis 1: Comparison: Portal Training and Home Visits vs Portal Training; Test type: Superiority; Group differences in expected 12 month c = -0.6, 95% CI 2-sided [-2.21 to 0.97]

4. Secondary Outcome: Hospitalizations
Description: Hospitalizations for asthma in the year before baseline to one year after baseline.
Time Frame: Hospitalizations for asthma in the year before baseline to one year after baseline
Population: rate per year
Measure: Least Squares Mean (95% Confidence Interval); unit: hospitalizations per year
Arm/Group | Portal Training and Home Visits | Portal Training
Number analyzed (Participants) | 151 | 150
hospitalizations per year | -1.19 [-1.56 to -0.80] | -0.66 [-1.02 to -0.30]
Statistical Analysis 1: Comparison: Portal Training and Home Visits vs Portal Training; Test type: Superiority; Group differences in expected 12 month c = -0.53, 95% CI 2-sided [-1.08 to -0.24]

5. Secondary Outcome: Prednisone Bursts
Description: new prescriptions of prednisone or increases in an already-prescribed dose for an asthma exacerbation measured at baseline and at one year.
Time Frame: bursts at baseline and at one year
Population: new prescriptions of prednisone or increases in an already-prescribed dose ("bursts") per year for an asthma exacerbation
Measure: Least Squares Mean (95% Confidence Interval); unit: bursts per year
Arm/Group | Portal Training and Home Visits | Portal Training
Number analyzed (Participants) | 151 | 150
bursts per year | -0.21 [-0.32 to -0.09] | -0.12 [-0.21 to -0.02]
Statistical Analysis 1: Comparison: Portal Training and Home Visits vs Portal Training; Test type: Superiority; Group differences in expected 12 month c = -0.09, 95% CI 2-sided [-0.24 to 0.06]

ADVERSE EVENTS:
Time Frame: One year
Description: Not different.
Arm/Group | Portal Training and Home Visits | Portal Training
All-Cause Mortality (participants affected / at risk) | 3/151 | 2/150
Serious Adverse Events (participants affected / at risk) | 49/151 | 63/150
Other Adverse Events (participants affected / at risk) | 14/151 | 18/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Portal Training and Home Visits (N=151) | Portal Training (N=150)
bronchospasm (Respiratory, thoracic and mediastinal disorders) | 40 | 42 — Uncontrolled asthma is an inclusion requirement. The vast number of adverse events are asthma-related exacerbations.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 4 — pneumonia
chest pain (Cardiac disorders) | 1 | 3
allergic reaction (Immune system disorders) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1
hypertension (Cardiac disorders) | 0 | 4
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
headache (Nervous system disorders) | 0 | 2
injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 | 3 — dog bite
bronchial infection (Respiratory, thoracic and mediastinal disorders) | 0 | 2
abdominal pain (Gastrointestinal disorders) | 0 | 1
GI reflux (Gastrointestinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
chest wall pain (Cardiac disorders) | 1 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
pain (General disorders) | 0 | 2
anaphlaxis (Immune system disorders) | 0 | 1
heart attack, myocardial infarction (Cardiac disorders) | 1 | 1
cardiac disorder (Cardiac disorders) | 0 | 1
colitis (Gastrointestinal disorders) | 0 | 1
heart failure (Cardiac disorders) | 1 | 0
hyperglycemia (Endocrine disorders) | 0 | 1
immune system disorder- Graves disease (Immune system disorders) | 0 | 1
oral pain (Gastrointestinal disorders) | 0 | 1
palpitations (Cardiac disorders) | 1 | 0
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Seizures (Nervous system disorders) | 0 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
sinusitis (Infections and infestations) | 1 | 0
upper respiratory infection (Infections and infestations) | 0 | 1
urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
penile infection (Infections and infestations) | 0 | 1
stroke (Nervous system disorders) | 2 | 1
anxiety (Psychiatric disorders) | 1 | 0
flu like symptoms (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Portal Training and Home Visits (N=151) | Portal Training (N=150)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 11 | 15
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
wheeze (Respiratory, thoracic and mediastinal disorders) | 1 | 1
bronchial infection (Infections and infestations) | 1 | 1
abdominal pain (Gastrointestinal disorders) | 0 | 1
acid reflux (Gastrointestinal disorders) | 0 | 1
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
chest pain (Cardiac disorders) | 1 | 0
dry eye (Eye disorders) | 1 | 0
short of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1
laryngitis (Infections and infestations) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/65/NCT02086565/Prot_SAP_000.pdf